CLINICAL TRIAL: NCT04882904
Title: Continuous Measurement of Activity in Patients With Muscle Pathology and in Control Subjects
Brief Title: Continuous Measurement of Activity in Patients With Muscle Pathology and in Control Subjects. ActiSLA Part.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: SYSNAV (Industry); Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Laurent Servais, Coordinator of reference center for neuromuscular diseases, Centre Hospitalier Universitaire de Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ActiLiège. ActiSLA part.
Record Dates: First submitted 2021-03-11; First posted 2021-05-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Actimyo; Accelerometry; Daily living
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: All patients undergo clinical evaluation and wear Actimyo device in daily living to evaluate their evolution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with ALS (Experimental): Patient with amyotrophic lateral sclerosis
  Interventions: Device: Actimyo°

INTERVENTIONS:
Device: Actimyo° — Actimyo° is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.

SUMMARY:
ActiSLA is a monocentric academic study. Patients with amyotrophic lateral sclerosis may be included on a voluntary basis. The investigators plan to include a group of approximately 20 patients with ALS.

The investigators have planned to assess patient every three months for a year. On each visit, participants will undergo a clinical examination with MRC sum score and Ashworth scores.

They will perform few tests ( 6-minutes walk test (6MWT), dynamometric measure, electromyography, Edinburgh Cognitive and Behavioural ALS Screen ) and will answer to some questionaires (dysphagia handicap scale, ALS-SFR-r).

After each visit, participants will wear Actimyo for one month daily.

ELIGIBILITY:
Inclusion Criteria:

* Clinically defined or probable diagnosis of ALS according to El Escorial criteria revised with Awaji's electro-diagnostic algorithm.
* Over 18 years old.
* Signed informed consent
* If patient on Riluzole, the dosage should be stable for 1 month and continued throughout the study period.

Exclusion Criteria:

* Patients with excessive cognitive disorders, limiting the understanding of task or with apparent communication difficulties hindering data collection.
* Any other previous or present pathology having an impact on motor function.
* Recent surgery or trauma (less than 6 months) in the upper or lower limbs.
* Prior neurological, endocrine, infectious, allergic, or chronic or acute inflammatory pathology in the three weeks preceding inclusion.
* Patients participating in an interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
95th centile of stride velocity | 1 year
  95th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter per second).
50th centile of stride velocity | 1 year
  50th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter per second).
95th centile of stride length | 1 year
  95th centile of stride length obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter).
50th centile of stride length | 1 year
  50th centile of stride length obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter).

SECONDARY OUTCOMES:
Upper limb function evolution in patient with ALS | 1 year
  Upper limb function assessed with a magneto-inertial sensor (Actimyo°) in real-life.

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Poleur, MD, Principal Investigator — CHR Citadelle-CHU liège
Locations (1):
- CHR Citadelle, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No